CLINICAL TRIAL: NCT06699394
Title: Teclistamab in Systemic AL Amyloidosis: a Multi-center Prospective Study
Brief Title: Prospective Study of Teclistamab in the Treatment of Systemic AL Amyloidosis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Jin Lu, MD, Dr, Peking University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023PHB319-001-03
Record Dates: First submitted 2024-11-18; First posted 2024-11-21 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: AL Amyloidosis
Keywords: teclistamab; complete hematological response
MeSH Terms: conditions — Immunoglobulin Light-chain Amyloidosis | interventions — Focal Adhesion Protein-Tyrosine Kinases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Group 1 (Other): Teclistamab monotherapy
  Interventions: Drug: Teclistamab (Tec)

INTERVENTIONS:
Drug: Teclistamab (Tec) — Teclistamab is administered subcutaneously with higher step-up doses (SUDs). Patients receive teclistamab with SUDs: 0.2 and 0.7 mg/kg and 1.5 mg/kg in Cycle 1 (2-4 days between doses). 3 mg/kg every 4 weeks will be used in subsequent cycles.

SUMMARY:
This study aims to evaluate the use of teclistamab in systemic AL amyloidosis and answer whether teclistamab can improve the rate of complete hematological response.

This is a single-arm, multi-center, prospective study. Participants will receive the single drug teclistamab, which the investigator deems the best choice.

DETAILED DESCRIPTION:
The treatment of amyloidosis should focus more on complete hematological response (CHR) and organ response rate. We hypothesize that teclistamab can deeply eliminate cloned plasma cells in AL patients, achieving a high proportion of complete hematological response.

In clinical practice, if daratumumab, bortezomib, and venetoclax (for patients with t(11;14)）have been used, the outcome is poor. Also, CHR is correlated with better clinical outcomes. In clinical routine practice, we use teclistamab, a more effective treatment to eliminate clonal plasma cells.

To further explore efficacy and safety, we designed this prospective study.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of systemic AL amyloidosis;
2. Patients must have received standard-of-care daratumumab, bortezomib, they do not have at least one organ response, and have not get complete hematological response;
3. Life expectancy greater than 12 weeks;
4. HGB ≥70g/L;
5. Blood oxygen saturation > 90%;
6. Total bilirubin (TBil) ≤3×upper limit of normal (ULN); aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤3.0×ULN;
7. Informed consent explained to, understood by and signed by the patient.

Exclusion Criteria:

1. Fulfill with the criteria of active multiple myeloma or active lymphoplasmacytic lymphoma.
2. Presence of other tumors which is/are in advanced malignant stage and has/have systemic metastasis;
3. Severe or persistent infection that cannot be effectively controlled;
4. Presence of severe autoimmune diseases or immunodeficiency disease;
5. Patients with active hepatitis B or hepatitis C ([HBVDNA+] or [HCVRNA+]);
6. Patients with HIV infection or syphilis infection;
7. Any situations that the researchers believe will increase the risks for the subject or affect the results of the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-03-29 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Complete hematological response | 3 months, 6 months
  Complete hematological response using ISA criteria

SECONDARY OUTCOMES:
Minimal residual disease | 3 months, 6 months
  Bone marrow minimal residual disease detected by multi-flow cytometry at the sensitivity of at least 10^-5.
Stringent dFLC response | 3 months, 6 months
  dFLC ≤ 10 mg/L
TRAE | 3 months, 6 months, 12 months
  Treatment realted adverse events
MOD-PFS | 12 months, 24 months
  The time from the beginning of treatment to death, clinical manifestation of end-stage cardiac or renal failure, or hematologic progression, whichever occurs first.
OS | 12 months, 24 months
  Overall survival
Renal Response | 3 months, 6 months, 12 months
  Renal Response according to ISA criteria
Cardiac Response | 3 months, 6 months, 12 months
  Cardiac Response according to ISA criteria
Hepatic Response | 3 months, 6 months, 12 months
  Hepatic Response according to ISA criteria

CONTACTS AND LOCATIONS:
Overall Officials: Jin Lu, M.D., Principal Investigator — Peking University People's Hospital
Locations (2):
- China (2):
  - Peking University Peoples Hospital, Beijing, Beijing Municipality
  - Fuxing Hospital affiliated to Capital Medical University, Beijing

IPD SHARING:
Plan to Share IPD: No